CLINICAL TRIAL: NCT05860959
Title: A Phase IV Longitudinal Study of SUBLOCADE (SUBUTEX Prolonged Release) Clinical Outcomes in Adults With Opioid Use Disorder (Opioid Dependence)
Brief Title: SUBLOCADE Long-term Outcomes
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INDV-6000-406
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder
Keywords: Medicine for Opioid Use Disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will provide the opportunity to generate data on the long-term use of SUBLOCADE under real-world conditions, and to observe enduring changes in lifestyle, health, and sociodemographic factors that are part of the recovery process. Long-term patterns of abstinence/opioid misuse as well as measures of participants' physical, psychological, social, and economic well-being will be monitored to better understand factors associated with recovery from opioid use disorder (OUD). Therefore, this study will observe participants up to a maximum of 4 years.

DETAILED DESCRIPTION:
This is a Phase IV, prospective, multicentre, multinational, open-label, real-world observational study in participants with current or a history of OUD/opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Is an adult ≥ 18 years of age who has signed the informed consent form
* Plans to receive additional SUBLOCADE injections and

  * Has initiated treatment for OUD/opioid dependence with SUBLOCADE within the last 3 months prior to Baseline Visit

    * OR
  * Has completed an Indivior SUBLOCADE study (eg, INDV-6000-401, INDV-6000-405) and has received the last dose of SUBLOCADE on that study within 3 months prior to Baseline Visit
* Is not currently participating in any clinical trial requiring medical intervention
* Is not currently using opioids to treat a diagnosis other than OUD/opioid dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants may enroll if they have initiated treatment with SUBLOCADE within 3 months prior to signing the informed consent form (ICF), or have completed an Indivior SUBLOCADE study (eg, INDV-6000-401, INDV-6000-405) and received their last dose of SUBLOCADE on the study within 3 months prior to signing the ICF, and plan to receive additional SUBLOCADE injections.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Participants achieving DSM-5 remission, early or sustained, (yes/no) while on initial SUBLOCADE treatment by 6 months and 1, 1.5, 2, 2.5, and 3 years from study Baseline | up to a maximum of 4 years
  * Definition of early remission: None of the criteria for OUD has been met for at least 3 months but for less than 12 months with the exception that Criterion 4 ("Craving, or a strong desire or urge to use opioids,") may be met.
  * Definition of sustained remission: None of the criteria for OUD has been met for at least 12 months with the exception that Criterion 4 ("Craving, or a strong desire or urge to use opioids,") may be met.

SECONDARY OUTCOMES:
Key Secondary: Participants with "no symptoms" or improving by ≥1 DSM-5 severity classification within the last 3 months (moderate to mild, or severe to mild or moderate) relative to study Baseline (yes/no) at Month 6 and Years 1, 2, and 3 | up to a maximum of 4 years
  DSM-5-Related
Among those starting SUBLOCADE within 3 months of study Baseline, time to achieve early remission for the first time while on initial SUBLOCADE treatment | up to a maximum of 4 years
  DSM-5-Related
Participants achieving DSM-5 sustained remission (yes/no) by 1, 1.5, 2, 2.5, and 3 years while on initial SUBLOCADE treatment | up to a maximum of 4 years
  DSM-5-Related
Time to achieve sustained remission for the first time while on initial SUBLOCADE treatment | up to a maximum of 4 years
  DSM-5-Related
Time to discontinuing initial SUBLOCADE treatment and the corresponding reasons for discontinuation, eg, resolution of OUD symptoms, safety concerns, treatment failure, or seeking alternative MOUD treatment | up to a maximum of 4 years
  MOUD Use and Retention
Participants switching from initial SUBLOCADE treatment to another MOUD (yes/no), and the corresponding reasons, eg, safety concerns, treatment failure, seeking alternative MOUD treatment | up to a maximum of 4 years
  MOUD Use and Retention
The overall treatment duration for participants who stop initial SUBLOCADE treatment as the result of resolution of OUD symptoms | up to a maximum of 4 years
  MOUD Use and Retention
Participants with any positive opioid use in the past month (yes/no) at Month 6 and Years 1, 2, and 3 while on initial SUBLOCADE treatment | up to a maximum of 4 years
  Illicit Opioid Use (Self-Reports)
Participants with opioid overdose requiring intervention (yes/no) while on initial SUBLOCADE treatment at least once during the first 6 months, and during Years 1, 2, and 3 | up to a maximum of 4 years
  Opioid Overdose Requiring Intervention

CONTACTS AND LOCATIONS:
Locations (49):
- United States (35):
  - ATP Clinical Research, Costa Mesa, California
  - Neighborhood Healthcare-Institute of Health, Escondido, California
  - Elevate Health and Wellness, Westport, Connecticut
  - United Research Institute, Hialeah, Florida
  - Zenith Clinical Research LLC, Hollywood, Florida
  - Jackson Health Community Center, Miami, Florida
  - G+C Research Group, Miami, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Collective Medical Research., Prairie Village, Kansas
  - Maine Health, Scarborough, Maine
  - Maryland Treatment Centers, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - THRYV Clinical Studies, Dearborn, Michigan
  - Vida Clinical Studies, Dearborn Heights, Michigan
  - Wayne State University Hospital, Detroit, Michigan
  - North Point Medical Center, Fair Haven, Michigan
  - SHMG Center for Integrative Medicine, Grand Rapids, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Psych Care Consultants, St Louis, Missouri
  - DENT Neurologic Institute, Amherst, New York
  - United Health Services, Binghamton, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Core Clinical Trials, North New Hyde Park, New York
  - Stuart Wasser Practice, Rockville Centre, New York
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - Pahl Pharmaceutical Professionals LLC, Oklahoma City, Oklahoma
  - Healing Comfort Clinic, LLC, Corvallis, Oregon
  - Thalia Medical Centre, Narberth, Pennsylvania
  - Charleston Pain and Rehabilitation Center, Charleston, South Carolina
  - Midlands Neurology, Columbia, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Alpine Research Organization, Clinton, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (4):
  - St Vincent's Hospital Melbourne, Fitzroy, Melbourne
  - John Hunter Hospital, Newcastle, New South Wales
  - Drug and Alcohol Services South Australia (DASSA), Stepney, South Australia
  - Turning Point, Richmond
- Canada (8):
  - Smart Clinic, Calgary, Alberta
  - Recovery Alberta, Edmonton, Alberta
  - Fraser Health Authority, Surrey, British Columbia
  - Dr. J.S. Dhillon Medicine Prof. Corp, Burlington, Ontario
  - The Stipley Clinic, Hamilton, Ontario
  - Brightshores Health System, Owen Sound, Ontario
  - Bluewater Rapid Assessment Addiction Medicine Clinic, Sarnia, Ontario
  - Comprehensive Treatment Clinic, Toronto, Ontario
- Sweden (2):
  - Linkoping University Hospital, Psychiatry Center, Linköping
  - Beroendecentrum, Stockholm

IPD SHARING:
Plan to Share IPD: No